CLINICAL TRIAL: NCT01545622
Title: Surgeon Compared to Nuclear Radiology Readers for Tc-99m Sestamibi Scans for Parathyroid Disease
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 104675
Record Dates: First submitted 2012-02-21; First posted 2012-03-07 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Parathyroid Disease
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze the findings of 30 surgeons and 30 nuclear radiologists of 61 individual thyroid scans. The goal is to determine if surgeons are more prone to making a definitive diagnosis based on a given scan than a nuclear radiologist. Accuracy of localization of the two groups will be analyzed. A secure website has been designed to which the physician will be able to login and view and rate the quality of each image and make a localizing diagnosis. Once they are finished, they will not be able to make any more changes, and their responses will be compared to the responses of their colleagues. The results will be analyzed to find if there is a significant variation in the ratings between the surgeons and the nuclear radiologists as to the quality, location, and number of parathyroid glands, if any, on the scans.

ELIGIBILITY:
Inclusion Criteria:

* Must be a surgeon or nuclear radiologist to be eligible read scans for this study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 surgeons and 30 nuclear radiologists.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Analyze the findings of individual thyroid scans | 1 day
  The results will be analyzed to find if there is a significant variation in the ratings between the surgeons and the nuclear radiologists as to the quality, location, and number of parathyroid glands, if any, on the scans.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Stack, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States